CLINICAL TRIAL: NCT06207799
Title: Pre-transplant Purging and Post-transplant MRD-guided Maintenance Therapy With Elranatamab in Patients With High-risk Multiple Myeloma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0448; NCI-2024-00110 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-01-05; First posted 2024-01-17 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Multiple Myeloma; Post-transplant MRD-guided Maintenance Therapy; Pre-transplant Purging
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; plerixafor; Melphalan; Busulfan; Granulocyte Colony-Stimulating Factor; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Elranatamab (Experimental): 1. Induction therapy - This is given to decrease the number of MM cells in the bone marrow.
  2. Purging - This is done to remove leftover MM cells after induction therapy.
  3. Stem cell mobilization - This is done to move stem cells from your bone marrow into the blood, so they can be collected for the autologous stem cell transplant.
  4. Conditioning therapy - This is given to help prepare the body to receive the stem cell transplant.
  5. Autologous stem cell transplant
  6. Maintenance therapy - This is given to help control the disease after the stem cell transplant.
  Interventions: Drug: Elranatamab; Drug: Lenalidomide; Drug: Plerixafor; Drug: Melphalan; Drug: Busulfan; Drug: G-CSF; Procedure: Stem cell transplant

INTERVENTIONS:
Drug: Elranatamab — Given by SC
  Other Names: PF-06863135
Drug: Lenalidomide — Given by PO
  Other Names: CC-5013; Revlimid™
Drug: Plerixafor — Given by SC
  Other Names: Mobozil
Drug: Melphalan — Given by IV
  Other Names: Alkeran®; Evomela
Drug: Busulfan — Given by PO
  Other Names: Busulfex™; Myleran®
Drug: G-CSF — Given by IV
Procedure: Stem cell transplant — Given by IV
  Other Names: Allogeneic stem cell transplant; Autologous stem cell transplant; Cord blood

SUMMARY:
To learn if giving elranatamab before and after an autologous stem cell transplant (ASTC) can help to control newly diagnosed, high-risk MM. An ASTC is a type of transplant in which a person's own stem cells are collected, preserved, and returned to them.

DETAILED DESCRIPTION:
Primary Objectives

* To determine the overall proportion of high-risk MM participants achieving sustained MRD-negative CR status after the completion of the treatment plan including in-vivo purging with elranatamab, auto-HCT, and post-transplant maintenance therapy. Sustained MRD-negativity is defined as MRD-negative status in two assessments, at least 1-year apart, without any MRD-positive status in between.
* To determine the proportion of patients with clonal plasma cell negative autograft collection in participants with high-risk MM.

Secondary Objectives

* To assess the impact of elranatamab on hematopoietic progenitor cell mobilization and collection yield.
* To determine the safety and tolerability of elranatamab plus lenalidomide maintenance therapy after auto-HCT.
* To detect the MRD-negative rate before auto-HCT with in-vivo purging using elranatamab.
* To detect the MRD-negative rate after auto-HCT.
* To determine overall response rates as defined by the International Myeloma Working Group (IMWG).
* To determine the PFS and OS with elranatamab plus lenalidomide maintenance therapy after auto-HCT in participants with high-risk NDMM.
* To determine the PFS and OS in participants with high-risk NDMM who discontinue maintenance therapy after achieving CR plus sustained MRD-negative status.
* To determine the PFS and OS with elranatamab plus lena

ELIGIBILITY:
Inclusion Criteria:

1. Transplant eligible patients with newly diagnosed multiple myeloma (NDMM).
2. High-risk multiple myeloma*
3. Participants with disease response ≥ PR to induction therapy
4. Age ≥ 18 and ≤ 75. Non-English-speaking participants are eligible.
5. Karnofsky performance status ≥70 (Appendix A).
6. Adequate liver function (total bilirubin ≤1.5X ULN; ALT ≤2.5 X ULN)
7. Estimated creatinine clearance ≥40 mL/min. Creatinine clearance may be calculated using Cockcroft-Gault, estimated glomerular filtration rate (Modification of Diet in Renal Disease [MDRD]), or Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula). *
8. Participant agrees to not donate blood while taking lenalidomide and for 28 days after stopping lenalidomide.
9. Participant agrees to enroll in the lenalidomide REMS program.
10. Women of child-bearing potential (WOCPB) must abstain from heterosexual intercourse or agree to use a contraceptive method that is highly effective (with a failure rate of <1% per year), preferably with low user dependency (as described in Appendix B), plus one additional effective method at least 28 days before starting therapy, during the intervention period, at least 28 days after the last dose of lenalidomide and at least 4 months after the last dose of elranatamab, and agrees not to donate eggs (ova, oocytes) for reproduction during this period. The investigator should evaluate the effectiveness of the contraceptive method in relation to the first dose of the study intervention. A WOCBP must have a negative highly sensitive serum pregnancy test (as required by local regulations) within 10-14 days and also within 24 hours before the first dose of the study intervention.

    Non Nonchildbearing potential is defined as follows (by other than medical reasons):
    * ≥ 45 years of age and has not had menses for >1 year.
    * Participants who have been amenorrhoeic for <2 years without a history of a hysterectomy and oophorectomy must have a follicle-stimulating hormone value in the postmenopausal range upon screening evaluation.
    * Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation.
11. Male participant agrees to contraceptive use that should be consistent with institutional guidelines regarding the methods of contraception for those participating in clinical studies.

    * Male participants are eligible to participate if they agree to the following during the intervention period and for 1 (for lenalidomide) to 4 (for elranatamab) months after the last dose of study treatment to allow for clearance of any altered sperm: - Refrain from donating sperm during treatment (including dose interruptions) and for 4 weeks after their last dose of lenalidomide and 4 months after the last dose of elranatamab.

    PLUS, either:
    * Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent. OR
    * Must agree to use contraception/barrier as detailed in Appendix B. *Definition of high-risk and ultra-high-risk MM15:
    * High-risk MM:

      o Presence of a high-risk chromosomal abnormality (HRCA) including: 17p13 deletion; t(4;14); t(14;16); t(14;20); Gain or amplification 1q by FISH.
    * Ultra-high-risk MM

      * Presence of ≥2 HRCA.

    Exclusion Criteria:

    • History of allergic reactions attributed to compounds of similar chemical or biologic composition to elranatamab or other agents used in study.

    • Drug interactions (Prohibited unless considered medically necessary):

    a. At projected clinical doses, TMDD (target mediated drug disposition) of elranatamab is expected. If concomitant medication alters target expression, it can potentially impact the PK of elranatamab. Drugs like anti-thymocyte globulin (ATG) can deplete T-cells and can potentially impact the PK of drugs targeting CD3. b. Elranatamab has been shown to increase T-cell activation and induce cytokine production (including IL-2, IL-6, IL-10, TNF-alpha and IFN-gamma). Cytokines have been shown to modulate expression of CYP enzymes and transporters, therefore, elranatamab can potentially affect CYP enzyme and transporter expression levels, and consequently modulate the clearance of concomitant medications that are substrates for these enzymes or transporters. When administering elranatamab, it is important to exercise caution with concomitant medications, especially those that are sensitive substrates of the cytochrome P450 (CYP) enzyme system and have a narrow therapeutic index. Increased exposure of CYP substrates is more likely to occur after the first dose of elranatamab on Day 1 and up to 14 days after the 32 mg dose on Day 4 and during and after CRS. Examples of such medications include cyclosporine. During this critical window, it's imperative to closely monitor the toxicity or concentrations of these concomitant drugs. If necessary, dose adjustments for these co-administered drugs should be considered to ensure patient safety. c. Cytochrome P450 (CYP) enzyme system is responsible for the metabolism of a vast number of drugs. Below are examples of drugs metabolized by specific CYP enzymes that could be impacted if elranatamab alters the activity or expression of these enzymes. Exercise caution when using these drugs: i. CYP2C9 substrates:

<!-- -->

1. - Warfarin
2. - Phenytoin
3. - Celecoxib
4. - Losartan ii. CYP3A4 substrates:

<!-- -->

1. - Statins: simvastatin, atorvastatin, lovastatin
2. - Calcineurin inhibitors: cyclosporine, tacrolimus
3. - Antiretroviral drugs: ritonavir, saquinavir, nelfinavir
4. - Benzodiazepines: diazepam, alprazolam
5. - Calcium channel blockers: nifedipine, verapamil, diltiazem
6. - Macrolide antibiotics: erythromycin, clarithromycin iii. CYP2D6 substrates:

<!-- -->

1. - Antipsychotics: aripiprazole, risperidone, haloperidol
2. - Tricyclic antidepressants: amitriptyline, nortriptyline, imipramine
3. - Beta-blockers: metoprolol, propranolol, carvedilol
4. - Codeine
5. - Tamoxifen iv. CYP1A2 substrates:

1. - Theophylline 2. - Fluvoxamine 3. - Clozapine v. CYP2C19 substrates:

1. - Omeprazole
2. - Citalopram
3. - Diazepam d. For participants on digoxin, monitor digoxin plasma levels periodically with the concomitant use of lenalidomide. Refer to lenalidomide USPI for additional information.

   • History of progressive disease at any time before starting maintenance.

   • Participants with non-secretory MM (no measurable disease on electrophoresis and immunofixation). Participants with a measurable disease on PET scan or bone marrow will be eligible.

   • Participants with Waldenströms macroglobulinemia.

   • Participants with POEMS syndrome.

   • Participants with smoldering MM (IMWG criteria)

   • Participants with plasma cell leukemia.

   • Participants with standard-risk MM.

   • Participants with relapsed and/or refractory MM.

   • Participant must not have presence of active renal condition (infection, requirement for dialysis or any other condition that could affect participant's safety). Participants with isolated proteinuria resulting from MM are eligible, provided they fulfil inclusion criteria.

   • Participant must not have current unstable liver or biliary disease defined by the presence of ascites, encephalopathy, coagulopathy, esophageal or gastric varices, persistent jaundice, or cirrhosis. Note: Stable non-cirrhotic chronic liver disease (including Gilbert's syndrome or asymptomatic gallstones) or hepatobiliary involvement of malignancy is acceptable if otherwise meets entry criteria.

   • Uncontrolled and active pulmonary disease.

   • Participant must not have used an investigational drug or approved systemic anti-myeloma therapy (including systemic steroids) within 14 days or five half-lives, whichever is shorter, preceding the first dose of study drug.

   • Participant must not have any evidence of active mucosal or internal bleeding.

   • Participant must not have an uncontrolled infection.

   • Participant must not have evidence of cardiovascular risk, including any of the following:
   * Evidence of current clinically significant uncontrolled arrhythmias, including clinically significant ECG abnormalities such as 2nd degree (Mobitz Type II) or 3rd degree atrioventricular (AV) block.
   * History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting or bypass grafting within three (3) months of screening.
   * Class III or IV heart failure as defined by the New York Heart Association functional classification system.16
   * Uncontrolled hypertension (blood pressure that remains above goal despite the concurrent use of three antihypertensive drug classes). • Participant must not have known HIV infection. • Participant must not have active Hepatitis B and/or C infection. • Participant must not have invasive malignancies other than disease under study, unless the second malignancy has been medically stable for at least 2 years and, in the opinion of the principal investigators, will not affect the evaluation of the effects of clinical trial treatments on the currently targeted malignancy. Participants with curatively treated non-melanoma skin cancer may be enrolled without a 2-year restriction. • Participants must not be pregnant or lactating. • Patients with cognitive impairments and/or any serious unstable pre-existing medical condition or psychiatric disorder that can interfere with safety or with obtaining informed consent or compliance with study procedures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Qaiser Bashir, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org